CLINICAL TRIAL: NCT00377793
Title: A Randomized, Double Blind, Parallel Group Study of Vardenafil Flexible Dose Versus Placebo in Males With Erectile Dysfunction and Their Female Partners Sexual Quality of Life. PARTNER II
Brief Title: Levitra (Vardenafil, BAY38-9456) Partner Satisfaction Study II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12146; EudraCT 2006-001228-37
Record Dates: First submitted 2006-09-08; First posted 2006-09-18 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Sexual Dysfunction; Male Erectile Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456)
  Arms: Arm 1
Drug: Placebo
  Arms: Arm 2

SUMMARY:
This trial is to provide additional important information on the impact of the treatment of the man its ED with vardenafil on partnership. This study is being run at up to 50 study centers in Europe and South Africa to evaluate the use of vardenafil in adult men with erectile dysfunction (often called impotence), and their female partner's sexual quality of life. Many men experience occasional erectile problems during their lives. However, when this becomes a continued problem, it can affect both the man and his female partner. The causes of erectile dysfunction are varied and may be due to physiological or emotional reasons. This study is designed to 1) study the effectiveness and safety of vardenafil, and 2) show whether treating a man its erectile dysfunction with vardenafil will improve his female partner its sexual quality of life. The second part (week 12) of the study (Educational program) a subgroup of subjects/couples, approximately 50% of the randomized subjects, will receive an educational program concerning ED in the from of a DVD.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 to 64 years
* Males with ED for more than six months, according to the NIH Consensus Statement (inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance)
* Stable heterosexual relationship for more than 6 months
* The subject must make at least four attempts at sexual intercourse
* Documented, dated, written Informed Consent Inclusion Criteria Partner
* Females 18 years, and older
* Stable, heterosexual relationship for more than 6 months with male ED subject
* Documented, dated, written Informed Consent
* Motivated to support treatment for male partner's ED
* Absence of significant sexual dysfunction as assessed by the total score on the FSFI16 > 23.55

Exclusion Criteria:

* Any unstable medical condition or substance abuse disorder that, in the opinion of the Investigator, is likely to affect the patient's ability to complete the study or precludes the patient's participation in the study
* Subjects who are taking nitrates or nitric oxide donors
* Subjects who are taking the following inhibitors of cytochrome P 450 CYP 3A4: very potent HIV protease inhibitors (ritonavir, indinavir), the anti-mycotic agents traconazole and ketoconazole (topical forms are allowed) or erythromycin
* Known hypersensitivity to vardenafil
* Presence of significant penile anatomical abnormalities (e.g. penile fibrosis or Peyronie's disease)
* History of retinitis pigmentosa
* Unstable angina pectoris
* Severe chronic or acute liver disease
* Premature ejaculator (defined as IELT < 2 minutes)
* Subjects who were taking alpha blockers
* Lost of vision of one eye because of NAION Exclusion Criteria Partner
* Presence of sexual dysfunction as assessed by the FSFI16 < 23.55
* Any unstable medical condition or substance abuse disorder that, in the opinion of the Investigator, is likely to affect the partner's ability to complete the study or precludes the partner's participation in the study

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2006-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Maintenance of erection in men with ED, Improvement of their female partners sexual quality of life | 12 weeks

SECONDARY OUTCOMES:
SEP3 at weeks 4, 12, 18, and 24 of treatment compared to placebo | 24 weeks
Additional Subject Diary questions at weeks 4, 12, 18, and 24, LOCF, and over entire treatment period compared to placebo | 24 weeks
Global confidence question (GCQ) at weeks 12, and 24 of treatment compared to placebo. IIEF, TSS, mSLQQ-QOL, Partnership questionnaire (PFB20) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (43):
- Belgium (5):
  - Bruxelles - Brussel
  - Genk
  - Leuven
  - Liège
  - Roeselare
- France (7):
  - La Rochelle
  - Lille
  - Lyon
  - Marseille
  - Mont-de-Marsan
  - Paris
  - Toulouse
- Germany (11):
  - Hamburg, Hamburg / 287
  - Hanover, Niedersachsen / 291
  - Brühl, Nordrhein-Westfalen / 325
  - Mülheim, Nordrhein-Westfalen / 481
  - Wuppertal, Nordrhein-Westfalen / 616
  - Bautzen, Sachsen / 313
  - Dresden, Sachsen / 313
  - Leipzig, Sachsen / 313
  - Leisnig, Sachsen / 313
  - Meißen, Sachsen / 313
  - Wahlstedt, Schleswig-Holstein / 306
- Italy (5):
  - Bergamo
  - Florence
  - Milan
  - Napoli
  - Roma
- Netherlands (4):
  - Arnhem
  - Deventer
  - Enschede
  - Nijverdal
- South Africa (4):
  - Bloemfontein, Free State
  - Johannesburg, Gauteng
  - Durban, KwaZulu-Natal
  - Newcastle, KwaZulu-Natal
- Spain (7):
  - Alicante, Alicante
  - Barcelona, Barcelona
  - La Roca del Vallès, Barcelona
  - Barcelona, Catalonia
  - Vigo, Pontevedra
  - San Cristóbal de La Laguna, Tenerife
  - Valencia, Valencia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/